CLINICAL TRIAL: NCT06523608
Title: Prediction of Decompensation and HCC Development in Patients With Advanced Chronic Liver Disease by the PLEASE and M10S20 Algorithms
Brief Title: Prediction of Decompensation and HCC Development in Advanced Chronic Liver Disease
Acronym: DETECT
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jonel Trebicka, Head of department of internal medicine B, University professor, Principal investigator, University Hospital Muenster
Other Study IDs: 2023-237-f-S
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Liver Diseases; Hepatocellular Carcinoma; Hepatocarcinoma; Advanced Chronic Liver Disease
MeSH Terms: conditions — Liver Diseases; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients in the control group are examined according to standard protocol (with a biannual follow-up) or more frequently when there is a development of decompensation or HCC.
  Interventions: Other: Standard survillance protocol
- Group with stratified surveillance: Patients in the study group will be stratified for the risk of decompensation/mortality and de novo-HCC-risk, based on the M10S20 ([Liver stiffness and MELD combined]) and PLEASE ([Platelet, Etiology, Age, Sex und Elastography]) scores.
  High-risk patients are allocated for a further CT/MRI examination and an AFP examination to exclude HCC and receive another appointment for a hospital visit within 3 months.
  Low-risk patients receive an appointment in one year.
  Interventions: Other: Stratified survillance protocol

INTERVENTIONS:
Other: Standard survillance protocol — Patients will be followed every 6 months. They will undergo at each visit an ultrasound examination including liver stiffness and a routine blood test, including AFP. Other examinations are carried out according to the standard of medical care. Blood, urine and stool tests as well as instrumental diagnostics such as duplex ultrasound, computer tomography, MR-tomography, endoscopies, bone marrow punctures, elastographies, TIPS implantations, operations, etc. will be performed as part of the usual diagnostic clarification.
  Groups: Control group
Other: Stratified survillance protocol — Based on PLEASE and M10LS20 scores, patients will be followed every 3 or 12 months. Low-risk patients will be followed once per year, and high-risk patients every 3 months.
  They will undergo at each visit an ultrasound examination including liver stiffness and a routine blood test, including AFP. Other examinations are carried out according to the standard of medical care. Blood, urine and stool tests as well as instrumental diagnostics such as duplex ultrasound, computer tomography, MR-tomography, endoscopies, bone marrow punctures, elastographies, TIPS implantations, operations, etc. will be performed as part of the usual diagnostic clarification.
  Groups: Group with stratified surveillance

SUMMARY:
The aim of this observational study is to predict the short- and long-term development of acute severe disease events, de novo hepatocarcinoma (HCC) and mortality in patients with advanced chronic liver disease using the M10S20 (Liver stiffness and Model for End-Stage Liver Disease Score [MELD] combined) and PLEASE (Platelet, Etiology, Age, Sex und Elastography) scores, as well as the validation of the cost-effectiveness of the algorithm.

Patients in this study are randomly divided into two groups:

* Control group: patients are examined according to the current clinical standard protocol (biannual follow-up).
* Stratified surveillance program:

  * High-risk patients will receive an appointment for a hospital visit every 3 months.
  * Low-risk patients could receive an appointment in one year. When necessary, if decompensation develops or HCC occurs, patients could be followed-up more frequently.

DETAILED DESCRIPTION:
Patients who are hospitalized with advanced chronic liver disease are randomly divided into two groups.

Patients in the control group are examined according to the current clinical standard protocol (biannual follow-up) or more frequently when decompensation or HCC develops.

Patients in the study group will be stratified for the risk of decompensation/mortality and de novo-HCC-risk, based on the M10S20 ([Liver stiffness and MELD combined]) and PLEASE ([Platelet, Etiology, Age, Sex und Elastography]) scores.

High-risk patients will be allocated for a further computer tomography (CT) or magnetic resonance imaging (MRI) examination and an alpha-fetoprotein (AFP) examination to exclude HCC and receive another appointment for a hospital visit within 3 months.

Low-risk patients could receive an appointment in one year. Patients in both arms, either outpatient or inpatient, will undergo at each visit an ultrasound examination with liver stiffness measurement and a routine blood test. Other examinations will be carried out according to standard medical care. Blood, urine and stool tests as well as instrumental diagnostics such as duplex ultrasound, CT, MRI, endoscopies, bone marrow punctures, elastographies, transjugular intrahepatic portosystemic shunt (TIPS) implantations, operations, etc. will be performed as part of the usual diagnostic clarification.

Hepatic encephalopathy is a decompensation event that will be diagnosed based on the West-Haven criteria, the number-connection test, the flicker frequency analysis and electroencephalogram. Written consent is required for every admitted patient. Data protection concept: When a patient is enrolled in the study, a center-specific study ID is first assigned for the purpose of pseudonymization.

The data collected is documented in an Excel spreadsheet. The assignment of the center-specific study ID to the respective patient is only possible for the respective investigator (Prof. Dr. Trebicka) and his staff (study nurse). For statistical evaluations, an analysis-specific data table will be created, which can be processed with an appropriate statistics program.

Patients cannot be identified with the data collected and the scientific research that derives from it.

ELIGIBILITY:
Inclusion Criteria:

* The patient admitted/referred to study center is hospitalized or is an outpatient with advanced chronic liver disease (based on the BAVENO criteria)

Exclusion Criteria:

* Pregnancy
* Age <18
* Evidence of current malignancy except for non-melanocytic skin cancer
* Presence or history of severe extra-hepatic diseases (e.g., chronic renal failure requiring hemodialysis, severe heart disease (New York Heart Association (NYHA) > II); severe chronic pulmonary disease (Global Initiative for Chronic Obstructive Lung Disease (GOLD) > III), severe neurological and psychiatric disorders).
* Human Immunodeficiency Virus (HIV) positive patients.
* Previous liver or other transplantation.
* Patients who decline to participate or who cannot provide prior written informed consent and when there is documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent.
* Physician's denial (e.g. the investigator considers that the patient will not follow the protocol scheduled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients should be included in the study if they are hospitalized with suspected chronic liver liver disease of viral and/or steatotic origin.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years
  All-cause mortality rate and liver-related mortality rate
Liver transplantation | 2 years
  Incidence of liver transplantation during follow-up period and time until liver transplantation.

SECONDARY OUTCOMES:
De novo HCC | 2 years
  Prediction of the risk of de novo HCC in patients with advanced chronic liver disease, based on the stratified surveillance, which can lead to earlier detection and treatment.
Acute liver decompensations | 2 years
  The acute occurrence of one or more complications of chronic portal hypertension, such as in patients with liver cirrhosis, a stable condition can develop into an acute decompensation. There is as well a new syndrome in patients with liver cirrhosis, which is characterized by a significantly increased hospitalization and a short-term (28-day) mortality rate. This syndrome is known as acute-on-chronic liver liver failure (ACLF).
  Portal hypertension is the driving force behind acute decompensation, while in the course of further decompensation and development of ACLF, an increasing, severe systemic inflammatory reaction is added.
Therapy in patients who develop HCC during follow-up | 2 years
  Assesment in the electronic case report form of number and type of therapies used to treat HCC (liver ablation, liver resection, chemoembolization, radiation or systemic therapy) when the patients develop HCC during the follow-up period.
Analysis of cost-effectiveness of the new algorithm compared to the routine follow-up | 2 years
  This outcome will be measured using the Markov model, which compares effectiveness based on Quality-adjusted life-years (QALYs) to the costs of each algorithm.
Analysis of proteome and metabolome in patients included into the study | 2 years
  Extraction of 40 ml of blood (30ml EDTA blood and 10ml serum) will be taken at each visit to the patient in addition to the regular diagnostics.
  This blood samples will be used to measure inflammatory markers (e.g. cytokines), components of the extracellular matrix components (e.g. collagens, matrix metalloproteinases), markers of bacterial translocation (e.g. LPS).
Analysis of intestinal and circulating microbiome in patients included into the study | 2 years
  Extraction of 40 ml of blood (30ml EDTA blood and 10ml serum) will be performed at each visit to the patient in addition to the regular diagnostics.
  A measurement of metagenome and 16S rRNA sequencing analyses will be performed in blood as well in stool samples to determine the composition of the intestinal and circulating microbiome.
Influence of circulating immune cells in HCC development and progression | 2 years
  Extraction of 40 ml of blood (30ml EDTA blood and 10ml serum) will be performed at each visit to the patient in addition to the regular diagnostics.
  From these blood samples circulating immune cells will be isolated, in order to investigate their influence on the disease.
Influence of transcriptome and metagenome in HCC development and progression | 2 years
  Extraction 30ml EDTA blood for DNA analysis will be performed at each visit to the patient in addition to the regular diagnostics. DNA/RNA extraction is used for transcriptome and metagenome analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jonel Trebicka, Prof. Dr. med., Principal Investigator — Department of Internal Medicine B, University Hospital Muenster, Muenster, Germany; Jonel Trebicka, Prof. Dr. med., Principal Investigator — European Foundation for Study of Chronic Liver Failure, Barcelona, Spain; Jonel Trebicka, Prof. Dr. med., Principal Investigator — Department of Gastroenterology and Hepatology, Odense University Hospital, Denmark
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Franchis R; Baveno V Faculty. Revising consensus in portal hypertension: report of the Baveno V consensus workshop on methodology of diagnosis and therapy in portal hypertension. J Hepatol. 2010 Oct;53(4):762-8. doi: 10.1016/j.jhep.2010.06.004. Epub 2010 Jun 27. No abstract available. PMID 20638742
- [Background] Kamath PS, Wiesner RH, Malinchoc M, Kremers W, Therneau TM, Kosberg CL, D'Amico G, Dickson ER, Kim WR. A model to predict survival in patients with end-stage liver disease. Hepatology. 2001 Feb;33(2):464-70. doi: 10.1053/jhep.2001.22172. PMID 11172350
- [Background] Jansen C, Moller P, Meyer C, Kolbe CC, Bogs C, Pohlmann A, Schierwagen R, Praktiknjo M, Abdullah Z, Lehmann J, Thomas D, Strassburg CP, Latz E, Mueller S, Rossle M, Trebicka J. Increase in liver stiffness after transjugular intrahepatic portosystemic shunt is associated with inflammation and predicts mortality. Hepatology. 2018 Apr;67(4):1472-1484. doi: 10.1002/hep.29612. Epub 2018 Feb 20. PMID 29059466
- [Background] Praktiknjo M, Book M, Luetkens J, Pohlmann A, Meyer C, Thomas D, Jansen C, Feist A, Chang J, Grimm J, Lehmann J, Strassburg CP, Abraldes JG, Kukuk G, Trebicka J. Fat-free muscle mass in magnetic resonance imaging predicts acute-on-chronic liver failure and survival in decompensated cirrhosis. Hepatology. 2018 Mar;67(3):1014-1026. doi: 10.1002/hep.29602. Epub 2018 Jan 24. PMID 29059469
- [Background] Lehmann J, Praktiknjo M, Nielsen MJ, Schierwagen R, Meyer C, Thomas D, Violi F, Strassburg CP, Bendtsen F, Moller S, Krag A, Karsdal MA, Leeming DJ, Trebicka J. Collagen type IV remodelling gender-specifically predicts mortality in decompensated cirrhosis. Liver Int. 2019 May;39(5):885-893. doi: 10.1111/liv.14070. Epub 2019 Mar 7. PMID 30739387
- [Background] Luo X, Leanza J, Massie AB, Garonzik-Wang JM, Haugen CE, Gentry SE, Ottmann SE, Segev DL. MELD as a metric for survival benefit of liver transplantation. Am J Transplant. 2018 May;18(5):1231-1237. doi: 10.1111/ajt.14660. Epub 2018 Feb 19. PMID 29316310
- [Background] Jansen C, Bogs C, Verlinden W, Thiele M, Moller P, Gortzen J, Lehmann J, Praktiknjo M, Chang J, Krag A, Strassburg CP, Francque S, Trebicka J. Algorithm to rule out clinically significant portal hypertension combining Shear-wave elastography of liver and spleen: a prospective multicentre study. Gut. 2016 Jun;65(6):1057-8. doi: 10.1136/gutjnl-2016-311536. Epub 2016 Feb 19. No abstract available. PMID 26896458
- [Background] Herrmann E, de Ledinghen V, Cassinotto C, Chu WC, Leung VY, Ferraioli G, Filice C, Castera L, Vilgrain V, Ronot M, Dumortier J, Guibal A, Pol S, Trebicka J, Jansen C, Strassburg C, Zheng R, Zheng J, Francque S, Vanwolleghem T, Vonghia L, Manesis EK, Zoumpoulis P, Sporea I, Thiele M, Krag A, Cohen-Bacrie C, Criton A, Gay J, Deffieux T, Friedrich-Rust M. Assessment of biopsy-proven liver fibrosis by two-dimensional shear wave elastography: An individual patient data-based meta-analysis. Hepatology. 2018 Jan;67(1):260-272. doi: 10.1002/hep.29179. Epub 2017 Nov 15. PMID 28370257
- [Background] Castera L, Friedrich-Rust M, Loomba R. Noninvasive Assessment of Liver Disease in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 Apr;156(5):1264-1281.e4. doi: 10.1053/j.gastro.2018.12.036. Epub 2019 Jan 18. PMID 30660725
- [Background] Wang K, Lu X, Zhou H, Gao Y, Zheng J, Tong M, Wu C, Liu C, Huang L, Jiang T, Meng F, Lu Y, Ai H, Xie XY, Yin LP, Liang P, Tian J, Zheng R. Deep learning Radiomics of shear wave elastography significantly improved diagnostic performance for assessing liver fibrosis in chronic hepatitis B: a prospective multicentre study. Gut. 2019 Apr;68(4):729-741. doi: 10.1136/gutjnl-2018-316204. Epub 2018 May 5. PMID 29730602
- [Background] Procopet B, Berzigotti A, Abraldes JG, Turon F, Hernandez-Gea V, Garcia-Pagan JC, Bosch J. Real-time shear-wave elastography: applicability, reliability and accuracy for clinically significant portal hypertension. J Hepatol. 2015 May;62(5):1068-75. doi: 10.1016/j.jhep.2014.12.007. Epub 2014 Dec 13. PMID 25514554
- [Background] Elkrief L, Rautou PE, Ronot M, Lambert S, Dioguardi Burgio M, Francoz C, Plessier A, Durand F, Valla D, Lebrec D, Vilgrain V, Castera L. Prospective comparison of spleen and liver stiffness by using shear-wave and transient elastography for detection of portal hypertension in cirrhosis. Radiology. 2015 May;275(2):589-98. doi: 10.1148/radiol.14141210. Epub 2014 Nov 28. PMID 25469784
- [Background] Robic MA, Procopet B, Metivier S, Peron JM, Selves J, Vinel JP, Bureau C. Liver stiffness accurately predicts portal hypertension related complications in patients with chronic liver disease: a prospective study. J Hepatol. 2011 Nov;55(5):1017-24. doi: 10.1016/j.jhep.2011.01.051. Epub 2011 Feb 25. PMID 21354450
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Cassinotto C, Lapuyade B, Guiu B, Marraud des Grottes H, Piron L, Merrouche W, Irles-Depe M, Molinari N, De Ledinghen V. Agreement Between 2-Dimensional Shear Wave and Transient Elastography Values for Diagnosis of Advanced Chronic Liver Disease. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2971-2979.e3. doi: 10.1016/j.cgh.2020.04.034. Epub 2020 Apr 26. PMID 32348907
- [Background] Monteiro S, Grandt J, Uschner FE, Kimer N, Madsen JL, Schierwagen R, Klein S, Welsch C, Schafer L, Jansen C, Claria J, Alcaraz-Quiles J, Arroyo V, Moreau R, Fernandez J, Bendtsen F, Mehta G, Gluud LL, Moller S, Praktiknjo M, Trebicka J. Differential inflammasome activation predisposes to acute-on-chronic liver failure in human and experimental cirrhosis with and without previous decompensation. Gut. 2021 Feb;70(2):379-387. doi: 10.1136/gutjnl-2019-320170. Epub 2020 Apr 2. PMID 32241903
- [Background] Praktiknjo M, Monteiro S, Grandt J, Kimer N, Madsen JL, Werge MP, William P, Brol MJ, Turco L, Schierwagen R, Chang J, Klein S, Uschner FE, Welsch C, Moreau R, Schepis F, Bendtsen F, Gluud LL, Moller S, Trebicka J. Cardiodynamic state is associated with systemic inflammation and fatal acute-on-chronic liver failure. Liver Int. 2020 Jun;40(6):1457-1466. doi: 10.1111/liv.14433. Epub 2020 Mar 30. PMID 32162397
- [Background] Trebicka J, Amoros A, Pitarch C, Titos E, Alcaraz-Quiles J, Schierwagen R, Deulofeu C, Fernandez-Gomez J, Piano S, Caraceni P, Oettl K, Sola E, Laleman W, McNaughtan J, Mookerjee RP, Coenraad MJ, Welzel T, Steib C, Garcia R, Gustot T, Rodriguez Gandia MA, Banares R, Albillos A, Zeuzem S, Vargas V, Saliba F, Nevens F, Alessandria C, de Gottardi A, Zoller H, Gines P, Sauerbruch T, Gerbes A, Stauber RE, Bernardi M, Angeli P, Pavesi M, Moreau R, Claria J, Jalan R, Arroyo V. Addressing Profiles of Systemic Inflammation Across the Different Clinical Phenotypes of Acutely Decompensated Cirrhosis. Front Immunol. 2019 Mar 19;10:476. doi: 10.3389/fimmu.2019.00476. eCollection 2019. PMID 30941129
- [Background] Poynard T, Munteanu M, Luckina E, Perazzo H, Ngo Y, Royer L, Fedchuk L, Sattonnet F, Pais R, Lebray P, Rudler M, Thabut D, Ratziu V. Liver fibrosis evaluation using real-time shear wave elastography: applicability and diagnostic performance using methods without a gold standard. J Hepatol. 2013 May;58(5):928-35. doi: 10.1016/j.jhep.2012.12.021. Epub 2013 Jan 12. PMID 23321316
- [Background] European Association for Study of Liver; Asociacion Latinoamericana para el Estudio del Higado. EASL-ALEH Clinical Practice Guidelines: Non-invasive tests for evaluation of liver disease severity and prognosis. J Hepatol. 2015 Jul;63(1):237-64. doi: 10.1016/j.jhep.2015.04.006. Epub 2015 Apr 21. No abstract available. PMID 25911335
- [Background] Hamada K, Saitoh S, Nishino N, Fukushima D, Horikawa Y, Nishida S, Honda M. Shear wave elastography predicts hepatocellular carcinoma risk in hepatitis C patients after sustained virological response. PLoS One. 2018 Apr 19;13(4):e0195173. doi: 10.1371/journal.pone.0195173. eCollection 2018. PMID 29672518
- [Background] Praktiknjo M, Krabbe V, Pohlmann A, Sampels M, Jansen C, Meyer C, Strassburg CP, Trebicka J, Gonzalez Carmona MA. Evolution of nodule stiffness might predict response to local ablative therapy: A series of patients with hepatocellular carcinoma. PLoS One. 2018 Feb 14;13(2):e0192897. doi: 10.1371/journal.pone.0192897. eCollection 2018. PMID 29444164
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Background] Gu W, Hortlik H, Erasmus HP, Schaaf L, Zeleke Y, Uschner FE, Ferstl P, Schulz M, Peiffer KH, Queck A, Sauerbruch T, Brol MJ, Rohde G, Sanchez C, Moreau R, Arroyo V, Zeuzem S, Welsch C, Trebicka J. Trends and the course of liver cirrhosis and its complications in Germany: Nationwide population-based study (2005 to 2018). Lancet Reg Health Eur. 2021 Nov 4;12:100240. doi: 10.1016/j.lanepe.2021.100240. eCollection 2022 Jan. PMID 34901909
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Background] Desai A, Sandhu S, Lai JP, Sandhu DS. Hepatocellular carcinoma in non-cirrhotic liver: A comprehensive review. World J Hepatol. 2019 Jan 27;11(1):1-18. doi: 10.4254/wjh.v11.i1.1. PMID 30705715
- [Background] Stine JG, Wentworth BJ, Zimmet A, Rinella ME, Loomba R, Caldwell SH, Argo CK. Systematic review with meta-analysis: risk of hepatocellular carcinoma in non-alcoholic steatohepatitis without cirrhosis compared to other liver diseases. Aliment Pharmacol Ther. 2018 Oct;48(7):696-703. doi: 10.1111/apt.14937. Epub 2018 Aug 22. PMID 30136293
- [Background] Lee DH, Lee JM. Primary malignant tumours in the non-cirrhotic liver. Eur J Radiol. 2017 Oct;95:349-361. doi: 10.1016/j.ejrad.2017.08.030. Epub 2017 Aug 31. PMID 28987692
- [Background] Benhammou JN, Lin J, Aby ES, Markovic D, Raman SS, Lu DS, Tong MJ. Nonalcoholic fatty liver disease-related hepatocellular carcinoma growth rates and their clinical outcomes. Hepatoma Res. 2021;7:70. doi: 10.20517/2394-5079.2021.74. Epub 2021 Nov 5. PMID 34966854
- [Background] Tobari M, Hashimoto E, Taniai M, Kodama K, Kogiso T, Tokushige K, Yamamoto M, Takayoshi N, Satoshi K, Tatsuo A. The characteristics and risk factors of hepatocellular carcinoma in nonalcoholic fatty liver disease without cirrhosis. J Gastroenterol Hepatol. 2020 May;35(5):862-869. doi: 10.1111/jgh.14867. Epub 2019 Dec 3. PMID 31597206
- [Background] Jiao Y, Dong F, Wang H, Zhang L, Xu J, Zheng J, Fan H, Gan H, Chen L, Li M. Shear wave elastography imaging for detecting malignant lesions of the liver: a systematic review and pooled meta-analysis. Med Ultrason. 2017 Jan 31;19(1):16-22. doi: 10.11152/mu-925. PMID 28180192
- [Background] Trebicka J, Gu W, de Ledinghen V, Aube C, Krag A, Praktiknjo M, Castera L, Dumortier J, Bauer DJM, Friedrich-Rust M, Pol S, Grgurevic I, Zheng R, Francque S, Gottfriedova H, Mustapic S, Sporea I, Berzigotti A, Uschner FE, Simbrunner B, Ronot M, Cassinotto C, Kjaergaard M, Andrade F, Schulz M, Semmler G, Drinkovic IT, Chang J, Brol MJ, Rautou PE, Vanwolleghem T, Strassburg CP, Boursier J, Ferstl PG, Rasmussen DN, Reiberger T, Vilgrain V, Guibal A, Guillaud O, Zeuzem S, Vassord C, Lu X, Vonghia L, Senkerikova R, Popescu A, Margini C, Wang W, Thiele M, Jansen C. Two-dimensional shear wave elastography predicts survival in advanced chronic liver disease. Gut. 2022 Feb;71(2):402-414. doi: 10.1136/gutjnl-2020-323419. Epub 2021 Jan 21. PMID 33479052
- [Background] Dold L, Nielsen MJ, Praktiknjo M, Schwarze-Zander C, Boesecke C, Schierwagen R, Mohr R, Wasmuth JC, Jansen C, Bischoff J, Rockstroh JK, Karsdal MA, Spengler U, Trebicka J, Leeming DJ. Circulating levels of PRO-C3 reflect liver fibrosis and liver function in HIV positive patients receiving modern cART. PLoS One. 2019 Jul 11;14(7):e0219526. doi: 10.1371/journal.pone.0219526. eCollection 2019. PMID 31295293
- [Background] Huang Y, de Boer WB, Adams LA, MacQuillan G, Bulsara MK, Jeffrey GP. Image analysis of liver biopsy samples measures fibrosis and predicts clinical outcome. J Hepatol. 2014 Jul;61(1):22-7. doi: 10.1016/j.jhep.2014.02.031. Epub 2014 Mar 6. PMID 24607623
- [Background] Daniels SJ, Leeming DJ, Eslam M, Hashem AM, Nielsen MJ, Krag A, Karsdal MA, Grove JI, Neil Guha I, Kawaguchi T, Torimura T, McLeod D, Akiba J, Kaye P, de Boer B, Aithal GP, Adams LA, George J. ADAPT: An Algorithm Incorporating PRO-C3 Accurately Identifies Patients With NAFLD and Advanced Fibrosis. Hepatology. 2019 Mar;69(3):1075-1086. doi: 10.1002/hep.30163. PMID 30014517
- [Background] Praktiknjo M, Simon-Talero M, Romer J, Roccarina D, Martinez J, Lampichler K, Baiges A, Low G, Llop E, Maurer MH, Zipprich A, Triolo M, Maleux G, Fialla AD, Dam C, Vidal-Gonzalez J, Majumdar A, Picon C, Toth D, Darnell A, Abraldes JG, Lopez M, Jansen C, Chang J, Schierwagen R, Uschner F, Kukuk G, Meyer C, Thomas D, Wolter K, Strassburg CP, Laleman W, La Mura V, Ripoll C, Berzigotti A, Calleja JL, Tandon P, Hernandez-Gea V, Reiberger T, Albillos A, Tsochatzis EA, Krag A, Genesca J, Trebicka J; Baveno VI-SPSS group of the Baveno Cooperation. Total area of spontaneous portosystemic shunts independently predicts hepatic encephalopathy and mortality in liver cirrhosis. J Hepatol. 2020 Jun;72(6):1140-1150. doi: 10.1016/j.jhep.2019.12.021. Epub 2020 Jan 15. PMID 31954206
- [Background] Simon-Talero M, Roccarina D, Martinez J, Lampichler K, Baiges A, Low G, Llop E, Praktiknjo M, Maurer MH, Zipprich A, Triolo M, Vangrinsven G, Garcia-Martinez R, Dam A, Majumdar A, Picon C, Toth D, Darnell A, Abraldes JG, Lopez M, Kukuk G, Krag A, Banares R, Laleman W, La Mura V, Ripoll C, Berzigotti A, Trebicka J, Calleja JL, Tandon P, Hernandez-Gea V, Reiberger T, Albillos A, Tsochatzis EA, Augustin S, Genesca J; Baveno VI-SPSS group from the Baveno Cooperation. Association Between Portosystemic Shunts and Increased Complications and Mortality in Patients With Cirrhosis. Gastroenterology. 2018 May;154(6):1694-1705.e4. doi: 10.1053/j.gastro.2018.01.028. Epub 2018 Jan 31. PMID 29360462
- [Background] Claria J, Stauber RE, Coenraad MJ, Moreau R, Jalan R, Pavesi M, Amoros A, Titos E, Alcaraz-Quiles J, Oettl K, Morales-Ruiz M, Angeli P, Domenicali M, Alessandria C, Gerbes A, Wendon J, Nevens F, Trebicka J, Laleman W, Saliba F, Welzel TM, Albillos A, Gustot T, Benten D, Durand F, Gines P, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium and the European Foundation for the Study of Chronic Liver Failure (EF-CLIF). Systemic inflammation in decompensated cirrhosis: Characterization and role in acute-on-chronic liver failure. Hepatology. 2016 Oct;64(4):1249-64. doi: 10.1002/hep.28740. Epub 2016 Aug 25. PMID 27483394
- [Background] Alvarez-Silva C, Schierwagen R, Pohlmann A, Magdaleno F, Uschner FE, Ryan P, Vehreschild MJGT, Claria J, Latz E, Lelouvier B, Arumugam M, Trebicka J. Compartmentalization of Immune Response and Microbial Translocation in Decompensated Cirrhosis. Front Immunol. 2019 Feb 8;10:69. doi: 10.3389/fimmu.2019.00069. eCollection 2019. PMID 30800122
- [Background] Verlinden W, Francque S, Michielsen P, Vanwolleghem T. Successful antiviral treatment of chronic hepatitis C leads to a rapid decline of liver stiffness without an early effect on spleen stiffness. Hepatology. 2016 Nov;64(5):1809-1810. doi: 10.1002/hep.28610. Epub 2016 Jun 7. No abstract available. PMID 27118145
- [Background] Castera L, Foucher J, Bernard PH, Carvalho F, Allaix D, Merrouche W, Couzigou P, de Ledinghen V. Pitfalls of liver stiffness measurement: a 5-year prospective study of 13,369 examinations. Hepatology. 2010 Mar;51(3):828-35. doi: 10.1002/hep.23425. PMID 20063276